CLINICAL TRIAL: NCT00508417
Title: Malaria Incidence in Infants in Bancoumana, Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907198; 07-I-N198
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-02-11

CONDITIONS: Malaria Infection; Malaria Incidence; Anemia
Keywords: Malaria Incidence; Anemia; Clinical Malaria
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study, conducted by the Malaria Research and Training Center at the Faculty of Medicine in Bamako and the NIAID will measure the frequency of occurrence of malaria in infants in Bancoumana, Mali. Information from the study will help in planning trials of malaria vaccines.

Healthy children from 6 weeks to 6 months of age who live in the Bancoumana health area may be eligible for this study. Candidates are screened with a physical examination and blood tests.

Participating children are visited at home for a total of about 17 visits to see if they are well. They come to the clinic every month during the 7-month study for a clinical evaluation, including a blood sample obtained by finger prick to test for malaria. Some of the blood collected may be stored and used for research. Children who become sick with malaria are treated for the disease.

DETAILED DESCRIPTION:
This is an observational study to determine the burden of malaria in rural Malian infants. Infants will be identified during a village-wide census and at Expanded Program for Immunization (EPI) visits. After obtaining community consent, eligible infants' parents will be invited to bring infants to the clinic for screening. Enrolled infants will receive a baseline evaluation and monthly visits during the rainy season at which times they will receive interim evaluations and heel, toe, or finger pricks for determinations of hemoglobin, thick and thin blood films, malaria antibody titers (at first and last visit for each transmission season), and hemoglobin typing at one visit. Study subjects will also receive a weekly home visit to determine if they are well or ill. If ill or febrile at any visit, or if they present to the clinic for an unscheduled visit, subjects will receive a history and physical examination, heel, toe, or finger pricks for determinations of hemoglobin, thick and thin blood films, filter paper blood collection and an RDT for malaria. Diagnosis and treatment of malaria will be performed according to Mali National Malaria Control Program (NMCP) guidelines. Diagnosis and treatment of other conditions will be performed as determined by the treating clinician.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Infants at least six weeks to less than 7 months of age at enrollment
  2. Known residents of the Bancoumana health area
  3. Good general health as determined by clinical exam
  4. Available for the 6-7 months duration of the trial
  5. Willingness to participate as evidenced by signing of the informed consent or fingerprinting by the parent or guardian

EXCLUSION CRITERIA:

1. Social, behavioral, cognitive, or psychiatric condition that in the opinion of the investigator affects the ability of the volunteer or the parent/legal guardian to understand and cooperate with the study protocol
2. Participation in an investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing
3. Infant born to mother with known or suspected HIV/AIDS as determined by the clinician

Ages: 6 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2007-07-24; Study Completion 2011-02-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), 9000 Rockville Pi, Bethesda, Maryland, United States

REFERENCES:
- [Background] Duflo B, Balique H, Ranque P, Diallo AN, Brucker G, Alavi H, Prescott N. [Estimation of the impact of the principal diseases in rural Mali]. Rev Epidemiol Sante Publique. 1986;34(6):405-18. French. PMID 3105007
- [Background] Wagner G, Koram K, McGuinness D, Bennett S, Nkrumah F, Riley E. High incidence of asymptomatic malara infections in a birth cohort of children less than one year of age in Ghana, detected by multicopy gene polymerase chain reaction. Am J Trop Med Hyg. 1998 Jul;59(1):115-23. doi: 10.4269/ajtmh.1998.59.115. PMID 9684638
- [Background] Moody AH, Chiodini PL. Non-microscopic method for malaria diagnosis using OptiMAL IT, a second-generation dipstick for malaria pLDH antigen detection. Br J Biomed Sci. 2002;59(4):228-31. doi: 10.1080/09674845.2002.11783665. PMID 12572958